

Approved by the Nemours IRB:

IRB# JAX: 332965

Valid from: 02/05/2016 through 02/04/2017

Abbreviated Study Title: MICT

## **NEMOURS**

## ADOLESCENT ASSENT FORM FOR YOUTH AGES 12-17 for the Asthma Research Study (revision date 09/23/2013)

## Title of Study: Use of Mobile Devices and the Internet to Streamline an Asthma Clinical Trial

I have had the study explained to me. I have been given a chance to ask questions. By answering the question below, I am saying whether or not I want to be in the study.

What is your decision about participating in this study called "Use of Mobile Devices and the Internet to Streamline an Asthma Clinical Trial"?

| | Yes, I want to participate in this study. |
|---|---|
| | No, I do not want to participate in this study. |
| Please type your first name in the box: This is your electronic signature. | |
| Please type your last name in the box: | |